CLINICAL TRIAL: NCT02778984
Title: Facial Mask Tightness: A Comparative Study
Acronym: EMAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: I15035
Record Dates: First submitted 2016-05-13; First posted 2016-05-20 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2017-05

CONDITIONS: Anesthesia
Keywords: Anesthesia; facial mask

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard face masks (Active Comparator): The standard mask is used in usual care
  Interventions: Other: standard mask
- QuadraLite face masks (Experimental): This study will compare tightness of 2 face masks during preoxygenation and after induction of anesthesia with propofol, sufentanil and rocuronium. During preoxygenation, a 10 l.min-1 fresh gas flow and 8 cm H2O PEEP will be applied. After induction of anesthesia, patients will receive pressure-controlled ventilation (fresh gaz flow 3 L.min-1, pressure set to obtain a 7 ml.kg-1 ideal body weight, 10 cpm, peep 5 cm H2O).
  Interventions: Device: QuadraLite masks

INTERVENTIONS:
Device: QuadraLite masks — The intervention is identical in the two group
  Arms: QuadraLite face masks
Other: standard mask
  Arms: standard face masks

SUMMARY:
A correct preoxygenation can be obtained after a 3min delay of calm ventilation through a tight mask thereafter mask is used to make the patient breathing before intubation. Most tight masks are actually sold but they have never been compared in studies. The aim of this study is to compare air leaks with standard facial mask and QuadraLite masks during preoxygenation and induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* edentulous patients
* age > 55 years

Exclusion Criteria:

* pregnancy or breast-feeding, patients on tutelage or guardianship
* patient unable to understand the protocol
* anesthesia in emergency or with full stomach

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
significant leakage (ie greater than 20% of the current volume) between QuadraLite® mask and facial mask | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No